CLINICAL TRIAL: NCT00170508
Title: In Depth Immunologic Studies in Healthy Young Adults Who Receive The Standard Dose Fluzone® (15mcgHA/Virus Strain) Trivalent Inactivated Influenza Virus Vaccine
Brief Title: Young Adult Influenza Vaccine Immunogenicity Substudy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 05-0055; Influenza CVD 12000
Record Dates: First submitted 2005-09-09; First posted 2005-09-15 (Estimated); Last update posted 2013-08-23 (Estimated); Status verified 2011-07

CONDITIONS: Influenza
Keywords: Influenza, sub-study
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

INTERVENTIONS:
Biological: Fluzone®

SUMMARY:
This is a complimentary study to an elderly influenza study. Subjects 18-40 will receive a single dose flu vaccine and be evaluated for humoral and cell mediated immunity to influenza antigens.

DETAILED DESCRIPTION:
The goals of this study are to provide in depth humoral and cellular immune responses to the standard-dose trivalent SV influenza virus vaccine containing 15 pg HA of each virus strain in healthy young adults. Serum samples will be submitted for the following analysis: measurement of serum anti-HA (hemagglutinin) IgG and IgA antibodies by ELISA, IgG antibody subclasses, IgG and IgA Avidity, Virus neutralizing functional assay, HAI antibody titer. Peripheral blood mononuclear cells (PBMC) isolated from these subjects will be evaluated for the following: "central" (TCM) and "effector" (TEM) memory T cell responses, including their proliferative responses and cytokine production profiles by flow cytometry, IFN-7 production by ELISPOT, following specific antigenic stimulation. Serum samples will be submitted for the following analysis: measurement ex vivo of the frequency of circulating influenza-specificT cells by using commercially available MHC/tetramers and/or MHC/pentamers and flow cytometry, role of regulatory T cells in the modulation of influenza responses in young adults. Fifteen healthy young adult subjects, age 18-40 years, inclusive, will be recruited from the general population to be enrolled in this study. No randomization or masking procedures will be used. All eligible subjects will be administered one intramuscular (IM) injection of the same FDA approved standard-dose (15 mcg HA per strain) trivalent inactivated influenza vaccine, 2004-2005 season, and key humoral and cell-mediated immunity (CMI) responses will be compared to those of elderly subjects enrolled under DMID 05-0028. On both Day 0 (pre-vaccination) and day 28 (post-vaccination), an 100 ml volume of whole blood will be obtained for a complete blood count (CBC) with differential and to isolate and cryopreserve serum and PBMCs. This study will evaluate key humoral and cell-mediated immunity (CMI) responses in healthy young adults to establish a baseline immune response which will be used to evaluate changes associated with immunosenescence. This study is linked to DMID protocol 05-0028.

ELIGIBILITY:
Inclusion Criteria:

1. Male or nonpregnant female (as indicated by a negative urine pregnancy test immediately prior to vaccine administration) between the ages of 18 and 40 years, inclusive.
2. Women of childbearing potential who are at risk of becoming pregnant must agree to practice adequate contraception (i.e., barrier method, abstinence, and licensed hormonal methods) for the entire study period (28 days).
3. In good health, as determined by medical history and a targeted physical examination, if necessary.
4. Able to understand and comply with planned study procedures.
5. Able to provide informed consent and be available for all study visits.

Exclusion Criteria:

1. Has a known allergy to eggs or other components of the vaccine.
2. Has a positive urine pregnancy test at screening or prior to vaccination (if female), is lactating, or has the intention to become pregnant within 3 months of enrollment in this study.
3. Is undergoing immunosuppression as a result of an underlying illness or treatment.
4. Has an active neoplastic disease or a history of any hematologic malignancy.
5. Is using oral or parenteral steroids, high-dose inhaled steroids (>800 mcg/day of beclomethasone dipropionate or equivalent) or other immunosuppressive or cytotoxic drugs.
6. Has a history of receiving immunoglobulin or other blood product within the 3 months prior to enrollment in this study.
7. Has received any other licensed vaccines within 2 weeks (for inactivated vaccines) or 4 weeks (for live vaccines) prior to enrollment in this study.
8. Has an acute or chronic medical condition that, in the opinion of the investigator, would render vaccination unsafe or would interfere with the evaluation of responses (this includes, but is not limited to: known chronic liver disease, significant renal disease, unstable or progressive neurological disorders, diabetes mellitus, and transplant recipients).
9. Has a history of severe reactions following immunization with contemporary influenza virus vaccines.
10. Has an acute illness, including an oral temperature greater than 100.4 degrees F, within one week of vaccination.
11. Received an experimental vaccine or medication within 1 month prior to enrollment in this study, or expects to receive an experimental vaccine, medication, or blood product during the 4 week study period.
12. Has any condition that would place the volunteer at an unacceptable risk of injury or any condition that in the opinion of the investigator may compromise the safety of the volunteer or integrity of the study.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2005-06; Primary Completion 2005-08 (Actual); Study Completion 2005-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Maryland Baltimore, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Chen WH, Cross AS, Edelman R, Sztein MB, Blackwelder WC, Pasetti MF. Antibody and Th1-type cell-mediated immune responses in elderly and young adults immunized with the standard or a high dose influenza vaccine. Vaccine. 2011 Apr 5;29(16):2865-73. doi: 10.1016/j.vaccine.2011.02.017. Epub 2011 Feb 23. PMID 21352939